CLINICAL TRIAL: NCT01001572
Title: A Multi-national, Multi-center, Double-blind, Randomized, Parallel Study Comparing the Efficacy and Safety of Valsartan/Amlodipine 160/5 mg to Valsartan 160 mg Alone in Patients With Mild to Moderate Essential Hypertension Not Adequately Controlled With Valsartan 160 mg Monotherapy
Brief Title: Efficacy and Safety of Valsartan/Amlodipine in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2317
Record Dates: First submitted 2009-10-15; First posted 2009-10-26 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Essential Hypertension
Keywords: Blood pressure; hypertension; Exforge; valsartan/amlodipine
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Valsartan; Amlodipine; Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Valsartan 160 mg (Active Comparator): One capsule Valsartan 160 mg and 1 tablet placebo to Valsartan/Amlodipine taken orally once daily at approximately 9:00 AM for 8 weeks
  Interventions: Drug: Valsartan 160 mg; Drug: Placebo
- Valsartan/amlodipine 160/5 mg (Experimental): One film-coated tablet Valsartan/amlodipine 160/5 mg and 1 capsule Placebo to Valsartan taken orally once daily at approximately 9:00 AM for 8 weeks
  Interventions: Drug: Valsartan/amlodipine 160/5 mg; Drug: Placebo
- Single-Blind Run-In Valsartan 160 mg (Other): Single-Blind Run-In treatment with one capsule Valsartan 160 mg taken orally once daily at approximately 9:00 AM for 4 weeks.
  Interventions: Drug: Valsartan 160 mg

INTERVENTIONS:
Drug: Valsartan/amlodipine 160/5 mg — Valsartan/amlodipine 160/5mg film coated tablets taken orally once daily.
  Other Names: Exforge® 160/5mg
  Arms: Valsartan/amlodipine 160/5 mg
Drug: Valsartan 160 mg — Valsartan 160 mg capsule taken orally once daily.
  Other Names: Diovan® 160mg
  Arms: Single-Blind Run-In Valsartan 160 mg; Valsartan 160 mg
Drug: Placebo — 1 capsule or tablet taken orally once daily
  Arms: Valsartan 160 mg; Valsartan/amlodipine 160/5 mg

SUMMARY:
This study assessed the efficacy and safety of the valsartan/amlodipine 160/5 mg single-pill combination in patients with uncomplicated essential hypertension not adequately controlled (MSDBP ≥90 mmHg and <110 mmHg) on valsartan 160 mg alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent
* Male or female ages 18 or older and less than 86 years
* Diagnosed as having essential diastolic hypertension, as follows:

  * Visit 2/Single-blind run-in entry, all participants MUST have a MSDBP ≥ 95 mmHg and < 100 mmHg
  * At Visit 3/Core double-blind treatment period entry, all patients MUST have a MSDBP >=90 mmHg and <110 mmHg

Exclusion Criteria:

* Severe hypertension
* Evidence of secondary form of hypertension (coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma or polycystic kidney disease )
* Malignant hypertension
* Administration of any agent indicated for the treatment of hypertension after Visit 1
* Known moderate or malignant retinopathy.
* Known or suspected contraindications, including history of allergy or hypersensitivity to Angiotensin II Receptor Blockers (ARBs), Calcium Channel Blockers (CCBs), or to drugs with similar chemical structures
* History of hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack, myocardial infarction or all types of revascularization, angina pectoris of any type, including unstable angina
* History of heart failure Grade II-IV according to New York Heart Association (NYHA) classification
* Second of third degree heart block regardless of the use of a pacemaker, concomitant potentially life-threatening arrhythmia or symptomatic arrhythmia

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH
Locations (2):
- Country not given (2):
  - Investigative site in Romainia
  - Novartis Investigative Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 932 participants were entered into the single-blind valsartan 160 mg arm. 278 participants were discontinued from the single-blind arm. 654 participants were randomized into the double-blind treatment phase; 329 to the Valsartan/amlodipine arm and 325 to the valsartan alone arm.
Groups:
- Single-Blind Run -In Valsartan 160 mg: Single-Blind Run-In treatment with one capsule Valsartan 160 mg taken orally once daily at approximately 9:00 AM for 4 weeks.
Period: Single-Blind Valsartan 160 mg
Arm/Group | Single-Blind Run -In Valsartan 160 mg | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Started | 932 | 0 (Participants did not enroll into this arm during single blind period.) | 0 (Participants did not enroll into this arm during single blind period.)
Completed | 654 | 0 | 0
Not Completed | 278 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Abnormal Test Procedure Result(s) | 96 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 7 | 0 | 0
Not completed — Abnormal Laboratory Value | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Administrative problems | 82 | 0 | 0
Not completed — Condition no longer requires study drug | 45 | 0 | 0
Period: Double-Blind Treatment Phase
Arm/Group | Single-Blind Run -In Valsartan 160 mg | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Started | 0 (This arm is only used for single blind period. So, no enrollment during double blind period.) | 329 | 325
Full Analysis Set (FAS) | 0 | 328 (One patient was excluded from full analysis set for having no post-baseline efficacy assessment.) | 323 (Two patients were excluded from full analysis set for having no post-baseline efficacy assessment.)
Completed | 0 | 319 | 306
Not Completed | 0 | 10 | 19
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 8 | 13
Not completed — Abnormal test procedure result(s) | 0 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg | Total
Number analyzed (Participants) | 328 | 323 | 651
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline Measures were based on the Full Analysis Set that excludes 3 participants for having no post-baseline efficacy assessment.
  years | 52.9 (9.47) | 53.1 (9.41) | 53.0 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 150 | 291
  Male | 187 | 173 | 360

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP) From Baseline to Week 8 Endpoint
Description: Three arterial blood pressure (BP) determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in the MSDBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from baseline in MSDBP was analyzed using an analysis of covariance model (ANCOVA) with treatment and center (pooled as appropriate) as factors and centered baseline MSDBP as a covariate.
Time Frame: Baseline and Week 8
Population: Full Analysis Set includes all randomized participants who had both baseline and at least one post-baseline efficacy measurement. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Number analyzed (Participants) | 328 | 323
mmHg | -10.3 (0.39) | -6.6 (0.40)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) From Baseline to Week 8 Endpoint
Description: Three arterial blood pressure (BP) determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in the MSSBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from baseline in MSSBP was analyzed using an analysis of covariance model (ANCOVA) with treatment and center (pooled as appropriate) as factors and centered baseline MSSBP as a covariate
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Number analyzed (Participants) | 328 | 323
mmHg | -14.9 (0.61) | -7.0 (0.61)

3. Secondary Outcome: Percentage of Participants With a Diastolic Blood Pressure Response at 8 Week Endpoint
Description: The percentage of participants with a Diastolic Blood Pressure Response defined as the percentage of participants with a Mean Sitting Diastolic Blood Pressure (MSDBP) < 90 mmHg or a >= 10 mmHg reduction from baseline.
Time Frame: Baseline and Week 8
Population: Full Analysis Set includes all randomized participants who had both baseline and at least one post-baseline efficacy measurement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Number analyzed (Participants) | 328 | 323
Percentage of Participants | 70.1 | 52.6

4. Secondary Outcome: Percentage of Participants With Diastolic Blood Pressure Control at 8 Week Endpoint
Description: The percentage of participants with Diastolic Blood Pressure Control defined as the percentage of participants with a Mean Sitting Diastolic Blood Pressure (MSDBP) < 90 mmHg.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Number analyzed (Participants) | 328 | 323
Percentage of Participants | 65.9 | 50.8

5. Secondary Outcome: Percentage of Participants With Overall Blood Pressure Control at 8 Week Endpoint
Description: The percentage of participants with Overall Blood Pressure Control defined as the percentage of participants with a Mean Sitting Systolic Blood Pressure (MSSBP)/Mean Sitting Diastolic Blood Pressure (MSDBP) < 140/90 mmHg.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Number analyzed (Participants) | 328 | 323
Percentage of Participants | 61.3 | 39.3

ADVERSE EVENTS:
Time Frame: Week 8
Description: Safety population included all randomized patients who received at least one dose of double-blind trial medication.
Arm/Group | Valsartan/Amlodipine 160/5 mg | Valsartan 160 mg
Serious Adverse Events (participants affected / at risk) | 0/329 | 1/325
Other Adverse Events (participants affected / at risk) | 0/329 | 0/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine 160/5 mg (N=329) | Valsartan 160 mg (N=325)
Uterine polyp (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.